CLINICAL TRIAL: NCT04108312
Title: Age-related Changes in Myeloarchitectonics Across Adulthood in Autism Spectrum Disorder
Status: Completed | Type: Observational
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Jiwandeep Kohli, Doctoral Research Fellow, San Diego State University
Other Study IDs: 11736
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Autism Spectrum Disorders
  Interventions: Diagnostic Test: Anatomical MRI Scan
- Typical Control
  Interventions: Diagnostic Test: Anatomical MRI Scan

INTERVENTIONS:
Diagnostic Test: Anatomical MRI Scan — T1-weighted (T1w) magnetization prepared rapid gradient echo (MPRAGE) sequence (TR=8.776 milliseconds, TE=3.656 milliseconds, flip angle=8°, matrix=320x320, 0.8mm3 resolution) and T2-weighted (T2w) CUBE sequence (TR=61.803 milliseconds, TE=3200 milliseconds, flip angle=8°, matrix=320x320, 0.8mm3 resolution)

SUMMARY:
There is increasing awareness in the Autism Spectrum Disorder (ASD) research field about the deficit of knowledge with regard to the neurobiological, cognitive, and behavioral changes that occur in adults with ASD across the later portion of the lifespan. Decline in motor skills and cognitive function in typical aging can have devastating impacts on an individual's ability to organize and maintain activities of daily living. While there is an overall lack of research on how these processes unfold across aging specifically in ASD, previous research findings of motor and cognitive deficits in young adults with ASD, localization of these functions to the anterior cerebral cortices, and trajectories of decline in typical aging indicate that motor skills and executive function are particularly at risk in the disorder in later life.

In vivo myeloarchitectonic mapping based on Magnetic Resonance Imaging (MRI) provides a unique view of gray matter structure and has the potential to elucidate abnormalities of local cortical connectivity. It has shown promise for the identification of biomarkers of disease pathogenesis in clinical studies, and it provides unique information beyond the cortical thickness measurements that have been employed in previous studies of ASD and typical aging. Myelin mapping may also be a more reliable index of neurobiological aging, given some questions about the accuracy of cortical thickness measurements. Given these properties, it may be a particularly informative measure in the context of potential accelerated decline in ASD. Intracortical myelin development and remodeling are protracted across the typical lifespan, with evidence of abnormal cortical myelination in other neuropsychiatric disorders, as well as in age-related mild cognitive impairment and dementia. In young adults with Autism Spectrum Disorder (ASD) myelin content is reduced in white matter and presumably in cortical gray matter as well. However, patterns of intracortical myelination have not yet been examined in ASD at any age leaving an important gap in the current knowledge base. With the added risk of demyelination associated with aging, older adults with ASD may be the most important population to examine as they may be doubly at risk of deficits in cortical myelination. Importantly, this could have knock-on effects on cognitive and motor functions in light of myelin's role in synaptic plasticity and maintenance of intracortical circuits.

The proposed fellowship project aims to bridge this gap in knowledge by investigating the age-related trajectory of intracortical myelin in middle aged to older adults with ASD and clarifying the spatial distribution of any abnormalities. Known heterogeneity in the clinical presentation and neurobiological phenotype across the autism spectrum poses a significant challenge in this research field. The proposed project includes innovative statistical approaches to help parse this heterogeneity. Intracortical myelin will be analyzed cross-sectionally using both group-wise and subject-specific approaches and with any findings confirmed with follow-up longitudinal data. This multifaceted approach will allow for a comprehensive characterization of myeloarchitectonics in adults with ASD, and also holds the potential to elucidate important links between brain structure and behavior in the disorder.

Specific Aims Aim 1: Determine if intracortical myelin content and rates of age-related change differ between individuals with ASD and age-matched control participants aged 40-65 years.

Hypothesis 1: Group-wise analysis will reveal decreased intracortical myelin content in ASD in association cortices of the frontal and parietal lobes.

Hypothesis 2: Subject-specific analyses may reveal spatial variability across individuals in the precise brain regions demonstrating abnormalities of intracortical myelination, but with frontal and parietal regions more frequently or more heavily affected.

Hypothesis 3: Both cross-sectional approaches will reveal a pattern of accelerated cortical demyelination with greater age in ASD.

Aim 2: Relate local myelin content measures to cognitive and behavioral abilities that are at-risk of decline during aging, including motor skills and executive functions.

Hypothesis 4: Age-related decline in domain-specific behavioral abilities will correlate with atypical patterns of intracortical myelination from Aim 1.

ELIGIBILITY:
Inclusion Criteria:

* ASD diagnoses to determine eligibility to participate in the study are made based on Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) criteria, supported by clinical interviews and the Autism Diagnostic Observation Schedule, Second Edition (ADOS-2)

Exclusion Criteria:

* Participants with a history of neurological (e.g. epilepsy, tuberous sclerosis) or genetic (e.g. fragile X, Rett syndrome) conditions other than ASD are excluded.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: San Diego County Community
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2015-05 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
Anatomical MRI Scan | Study Visit 2 - 1 hour scan session
  T1-weighted (T1w) magnetization prepared rapid gradient echo (MPRAGE) sequence (TR=8.776 milliseconds, TE=3.656 milliseconds, flip angle=8°, matrix=320x320, 0.8mm3 resolution) and T2-weighted (T2w) CUBE sequence (TR=61.803 milliseconds, TE=3200 milliseconds, flip angle=8°, matrix=320x320, 0.8mm3 resolution)

CONTACTS AND LOCATIONS:
Locations (1):
- San Diego State University, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No